CLINICAL TRIAL: NCT03392480
Title: Determination of the Association of Haptoglobin 2-2 With Delirium After Orthopedic Surgery
Brief Title: Association of Haptoglobin 2-2 With Postoperative Delirium
Status: Withdrawn | Type: Observational
Why Stopped: The research group cannot found time to do the project.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhiyi Zuo, Visiting Professor, Sun Yat-sen University
Other Study IDs: S2017-096-02
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum or plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult non-haptoglobin 2-2 group: Patients are 45 to 65 years old.
- Adult haptoglobin 2-2 group: Patients are 45 to 65 years old.
- Elder non-haptoglobin 2-2 group: Patients are elder than 65 years.
- Elder haptoglobin 2-2 group: Patients are elder than 65 years.

SUMMARY:
Patients with major orthopedic surgery will be recruited. Participants will be monitored for delirium after surgery. Participants' blood will be harvested for the determination of haptoglobin types, levels of oxidative stress and inflammation. Investigators will then analyze the data to see if haptoglobin 2-2 type is associated with an increased postoperative delirium, inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I to III class for major orthopedic surgery (hip or knee replacement or spinal surgery)
* No psychological and psychiatric history and presentation before surgery
* No major organ dysfunction or failure

Exclusion Criteria:

* Anemia (hemoglobin < 100 g/l) preoperatively.
* Requires > 4 units of allogeneic red blood cell transfusion during the surgery
* Using steroids or anti-psychological and anti-psychiatric drugs. A small dose of steroid for postoperative anti-nausea/vomiting is allowed and will not be considered as a indication for exclusion.
* Can not cooperate with the study
* History of bleeding
* BMI < 18 or > 30
* History of hemoglobin metabolism disorder

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusive criteria will be screened as possible candidates.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium incidence | From day 0 to up to 7 days after the surgery
  The incidence of delirium as assessed by intensive care unit-confusion assessment method will be determined.
Postoperative delirium duration | From day 0 to up to 7 days after the surgery
  The duration of delirium as assessed by intensive care unit-confusion assessment method will be determined.

SECONDARY OUTCOMES:
Oxidative stress level | Day 0 to day 2 after the surgery
  The level of malondialdehyde in the blood will be measured by ELISA.
Inflammation level | Day 0 to day 2 after the surgery
  The levels of interleukin 1beta and interleukin 6 in the blood will be assessed by ELISA.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Jishuitan hospital, Beijing
  - Chinese PLA general hospital, Beijing
  - Xinqiao hospital, Army military medical university, Chongqing
  - Daping Hospital, Army Military Medical University, Chongqing
  - the First Affiliated Hospital of Southern Medical University, Guangzhou
  - Third affiliated hospital of southern medical university, Guangzhou
  - shanghai Changzheng hospital, Naval Military Medical University, Shanghai
  - Shenyang general hospital of military region, Shenyang

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers